CLINICAL TRIAL: NCT01564212
Title: Quantitative Heat Loss With Laminar Air Flow
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 12-217
Record Dates: First submitted 2012-03-23; First posted 2012-03-27 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Healthy
Keywords: heat loss; laminar airflow; operating rooms
MeSH Terms: interventions — Surgical Drapes

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- standard airflow and forced air warming (Active Comparator): Subjects will lie on operating room bed with standard airflow and forced air warming.
  Interventions: Other: standard airflow with forced air warming.
- laminar airflow with surgical drapes (Active Comparator): Subjects will lie on operating room bed with laminar airflow device on and surgical drapes surrounding bed.
  Interventions: Other: laminar airflow with surgical drapes
- laminar aiflow with forced air warming (Active Comparator): Subjects will lie on operating room bed with laminar airflow on and warming forced air.
  Interventions: Other: laminar airflow with forced air warming
- standard airflow with surgical drapes (Active Comparator): Subjects will lie on operating room bed with standard airflow and surgical drapes surrounding bed.
  Interventions: Other: standard airflow with surgical drapes

INTERVENTIONS:
Other: standard airflow with forced air warming. — Subjects will lie on operating room bed with standard airflow and forced air warming.
  Arms: standard airflow and forced air warming
Other: laminar airflow with surgical drapes
  Other Names: Subjects will lie on operating room bed with laminar airflow and surgical drapes surrounding bed.
  Arms: laminar airflow with surgical drapes
Other: laminar airflow with forced air warming — Subjects will lie on operating room bed with laminar airflow and forced air warming.
  Arms: laminar aiflow with forced air warming
Other: standard airflow with surgical drapes — Subjects will lie on operating room bed with standard airflow on and surgical drapes surrounding bed.
  Arms: standard airflow with surgical drapes

SUMMARY:
With approval of the IRB at the Cleveland Clinic and written informed consent, the investigators propose to study up to 20 healthy volunteers in the protocol below as this will allow for drop-outs. As the investigators believe that 10 volunteers will provide sufficient power to detect clinically-meaningful differences between laminar air flow treatments.

The study has been designed to find out whether heat loss increases significantly in laminar air flow operating rooms. Furthermore the investigators will find out whether active warming minimizes this heat loss. Increased heat loss increases the amount of perioperative hypothermia. It has been shown that perioperative hypothermia is associated with severe complications such as an increased incidence of surgical wound infections. On the other hand laminar air flow is explicitly used to decrease air-borne infections. Our study results will help to optimize thermal management of orthopedic patients.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 45 years of age
* Healthy male and female volunteers
* ASA physical status I
* Capable and willing to provide written informed consent

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2012-03; Primary Completion 2017-02 (Actual); Study Completion 2017-02-23 (Actual)

PRIMARY OUTCOMES:
heat loss | 20 minutes
  Defining the within-volunteer difference in heat flux between laminar air flow 'on' and laminar air flow 'off' as the primary outcome of interest, we will use two linear regression models to perform analyses, respectively, for active warming and no active warming settings. Ambient temperature and relative humidity will be adjusted for within this linear model if they are not adequately balanced between the four experimental scenarios, on average (as determined by standard univariable summary statistics).

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Kurz, M.D., Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States